CLINICAL TRIAL: NCT01488513
Title: A Phase I, Open-label, Dose-Escalation, Safety, Pharmacokinetic and Pharmacodynamic Study of ABC294640 in Patients With Advanced Solid Tumors
Brief Title: ABC294640 in Treating Patients With Advanced Solid Tumors
Acronym: ABC-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Collaborators: Apogee Biotechnology Corporation (Industry); Medical University of South Carolina (Other); FDA Office of Orphan Products Development (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTO 101504; NCI -2011-02993 (Registry Identifier: CTRP(Clinical Trial Reporting Program)); G04102-00 (Other Grant/Funding Number: OOPD); R01FD004102-01 (FDA)
Record Dates: First submitted 2011-09-29; First posted 2011-12-08 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2015-08

CONDITIONS: Pancreatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: ABC294640; RedHill Biopharma, Ltd.; ABC-101; Medical University of South Carolina; Apogee Biotechnology Corporation
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 3-(4-chlorophenyl)-adamantane-1-carboxylic acid (pyridin-4-ylmethyl)amide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive sphingosine kinase-2 inhibitor ABC294640 PO BID on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sphingosine kinase-2 inhibitor ABC294640

INTERVENTIONS:
Drug: sphingosine kinase-2 inhibitor ABC294640 — Given PO Starting dose of ABC294640 250 mg once on day on Days 1-28 of each 28-day cycle. Subsequent cohort doses (if reached) are as follows: 250 BID, 500 BID, 750 BID, 1,000 BID, 1,500 BID, 2,000 BID, 2,500 BID
  Other Names: SK2 inhibitor ABC294640

SUMMARY:
This phase I trial studies the side effects and best dose of ABC294640 in treating patients with advanced solid tumors. ABC294640 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Please note that the FDA OOPD is participating as a funding source.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess safety and determine the maximum tolerated dose (MTD) and the dose limiting toxicities (DLT) of ABC294640 (sphingosine kinase-2 inhibitor ABC294640) in patients with solid organ tumors. (Part I) II. To assess the safety and tolerability of ABC294640 at the MTD in an expanded cohort of hepatocellular carcinoma (HCC) patients. (Part II)

SECONDARY OBJECTIVES:

I. To establish the dose of ABC294640 recommended for future phase II protocols. (Part I) II. To describe the pharmacokinetics of ABC294640 in patients with solid organ tumors. (Part I) III. To describe the effects of ABC294640 on plasma levels of sphingosine 1-phosphate in patients with solid organ tumors. (Part I) IV. To assess antitumor activity of ABC294640 in patients with solid organ tumors by objective radiographic assessment using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria. (Part I) V. To describe the pharmacokinetics of ABC294640 in HCC patients. (Part II) VI. To describe the effects of ABC294640 on plasma levels of sphingosine 1-phosphate in HCC patients. (Part II) VII. To assess antitumor activity of ABC294640 in HCC patients by objective radiographic assessment using RECIST 1.1 criteria. (Part II)

OUTLINE: This is a dose-escalation study.

Patients receive sphingosine kinase-2 inhibitor ABC294640 orally (PO) twice daily (BID) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up monthly for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* PART I:
* Patients with histologically confirmed solid organ carcinomas
* Tumor progression after receiving standard/approved chemotherapy or as first-line therapy for malignancies where there is no standard therapy
* One or more tumors measurable on computed tomography (CT) scan per RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of at least 3 months
* Age > 18 years
* Signed, written Institutional Review Board (IRB)-approved informed consent
* A negative pregnancy test (if female)
* Acceptable liver function:
* Bilirubin =< 3 times upper limit of normal (ULN) (Common Terminology Criteria for Adverse Events [CTCAE] Grade 2 baseline)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]), alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 3 x ULN (CTCAE Grade 1 baseline)
* Serum creatinine =< 1.5 X ULN (CTCAE Grade 1 baseline)
* Absolute neutrophil count >= 1000 cells/mm^3
* Acceptable hematologic status:
* Absolute neutrophil coun > 1000 cells/mm3
* Platelet count >= 75,000 (plt/mm^3) (CTCAE Grade 1 baseline)
* Hemoglobin >= 9 g/dL
* Acceptable blood sugar control:
* Fasting glucose value < 160 mg/dL (CTCAE Grade 1 baseline)
* Urinalysis: No clinically significant abnormalities
* Prothrombin time (PT) and partial thromboplastin time (PTT) =< 1.5 X ULN after correction of nutritional deficiencies that may contribute to prolonged PT/PTT
* For men and women of child-producing potential, willingness to use of effective contraceptive methods during the study; if female (or female partner of male subject), is either not of childbearing potential (defined as postmenopausal for >= 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or practicing 1 of the following medically acceptable methods of birth control and agrees to continue with the regimen throughout the duration of the study:
* Oral, implantable or injectable contraceptives for 3 consecutive months before the baseline/randomization visit
* Total abstinence from sexual intercourse (>= 1 complete menstrual cycle before the baseline/randomization visit)
* Intrauterine device (IUD)
* Double barrier method (condoms, sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* PART II:
* To be eligible for inclusion in Part II, patients must meet the eligibility for Part 1 as well as the following:
* Patients with histologically confirmed HCC for whom there is no standard/approved chemotherapy

Exclusion Criteria:

* New York Heart Association Class III or IV, cardiac disease, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG)
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Pregnant or nursing women; NOTE: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to study entry
* Unwillingness or inability to comply with procedures required in this protocol
* Known infection with human immunodeficiency virus (HIV)
* Serious nonmalignant disease (e.g., hydronephrosis, liver failure, or other conditions) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor
* Patients who are currently receiving any other investigational agent
* Patients who are receiving drugs that are sensitive substrates of CYP450 1A2, 3A4, 2C9, 2C19 or 2D6, or strong inhibitors or inducers of all major CYP450 isozymes that cannot be stopped at least 7 days or 5 half-lives (whichever is longer) before starting treatment with ABC294640 and either replaced with another appropriate medication or not given for the duration of the clinical study
* Patients who are currently taking Coumadin or Coumadin derivatives
* Patients who have received any antineoplastic therapy within 1 month of starting treatment with ABC294640 or who have not adequately recovered from side effects and toxicities of previous antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) defined as highest dose of ABC294640 at which 0 or 1 patient of 6 experiences a DLT. | Patients will be followed until the point in time when no more than 1 of 6 patients has a Dose Limiting Toxicity (DLT) in cycle 1, and expected 54 days.
  MTD defined as the highest dose at which 0 or 1 patient of 6 experiences a DLT. The DLT rate will be estimated with its 95% confidence interval.
Safety assessed using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0. | Weekly during course 1, bi-weekly for all subsequent courses, and at the end of treatment study-- expected to occur at an average of 6 months from study start.
  Assessed using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0. Adverse events (AEs) will be coded by body system and summary tables with incidence rates of adverse events will be generated. Descriptive statistics of AEs will be reported by doses and for subsets of patients with serious adverse events (SAEs), patients who discontinue due to AEs, and patients with related AEs.

SECONDARY OUTCOMES:
Pharmacodynamic parameters for sphingosine kinase-2 inhibitor ABC294640 | Days 1 and 28 of cycle 1 collected at prior to dose, 1, 2, 4, 8, 12, 24 hours post drug administration.
  Area under the drug concentration over time curve (AUC), maximum concentration, minimum concentration, and time to maximum concentration will be calculated for each subject.
Pharmacodynamic parameters for sphingosine kinase-2 inhibitor ABC294640 | Weekly during course 1, bi-weekly for all subsequent courses, and at the end of treatment study-- expected to occur at an average of 6 months from study start.
  Pharmacodynamic parameters for ABC294640 action will include measurement of plasma levels of S1P, including absolute concentration at each sampling time and chance from baseline concentration at each sampling time after drug administration.
Tumor response rate | Every 8 weeks till end of treatment study-- expected to occur at an average of 6 months from study start.
  All patients who have measureable disease according to RECIST 1.1, received at least one cycle of treatment, and have had disease re-evaluated will be included.

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States